CLINICAL TRIAL: NCT02499419
Title: Exercise Capacity Evaluation in Patients With Non-rheumatic Mitral Valve Prolapse (MVP)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0294-14-CTIL
Record Dates: First submitted 2014-10-27; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Mitral Valve Prolapse
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Healthy: Individuals without any known heart/ respiratory/ metabolic problems that might limit their exercise capacity
- Mild MVP: 0 or 1 of the following secondary risk factors: Mild MR Flail leaflet Left atrial diameter > 40 mm Atrial fibrillation Age ≥ 50
- Moderate MVP: 2 or more of the above secondary risk factors.
- Severe MVP: 1 or more of the following primary risk factors: EF < 50% MR ≥ moderate

SUMMARY:
Mitral valve prolapse (MVP) is a relatively common cardial problem in which one or more of the leaflets of the mitral valve prolapse during systole into the left atrium.

The disease is very heterogeneous and can vary from a benign disease with almost no impact on the patient's life to a severe cardiac problem with many complications and high mortality rate.

The purpose of the study is to see if the investigators can find a relation between the severity of the MVP to the exercise capacity of the patient. The investigators also want to see if they can find a difference between the exercise capacity of mild MVP patients and healthy people.

To evaluate the exercise capacity of the subjects the investigators use Cardiopulmonary Exercise Testing (CPET). CPET is probably the best known way to get a full picture of the subject's functions during exercise. By combining gas exchange monitoring and ECG during a controlled exercise in which the subject reaches maximal effort, the test gives information about the cardiac, the pulmonary and the metabolic functions of the subject. This information can help identify if there is a problem to perform exercise properly and more specifically if the limitation is due to a cardiac, pulmonary or metabolic problem.

DETAILED DESCRIPTION:
Mitral valve prolapse (MVP) is a relatively common cardial problem in which one or more of the leaflets of the mitral valve prolapse during systole into the left atrium.

The disease is very heterogeneous and can vary from a benign disease with almost no impact on the patient's life to a severe cardiac problem with many complications and high mortality rate .

The purpose of the study is to see if the investigators can find a relation between the severity of the MVP to the exercise capacity of the patient. The investigators also want to see if they can find a difference between the exercise capacity of mild MVP patients and healthy people.

To evaluate the exercise capacity of the subjects the investigators use Cardiopulmonary Exercise Testing (CPET). CPET is probably the best known way to get a full picture of the subject's functions during exercise. By combining gas exchange monitoring and ECG during a controlled exercise in which the subject reaches maximal effort, the test gives information about the cardiac, the pulmonary and the metabolic functions of the subject. This information can help identify if there is a problem to perform exercise properly and more specifically if the limitation is due to a cardiac, pulmonary or metabolic problem.

ELIGIBILITY:
Inclusion Criteria:

* MVP diagnosis
* Signing consent form (By parents if the patient is a minor)

Exclusion Criteria:

* Other congenital or acquired cardiac problems other than MVP.
* Patients with other diseases that can affect the exercise capacity.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People diagnosed with MVP and no other cardiac problems.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-10 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity as a measure of maximal oxygen uptake (VO2max), Anaerobic threshold and work efficiency | Within 30 days after the CPET test

SECONDARY OUTCOMES:
Exercise capacity limitation as a measure of the O2-pulse, heart rate, blood pressure, blood saturation, ECG and the ventilatory equivalents. | Within 30 days after the CPET test
The severity of the MVP as a measure of the mitral regurgitation, ejection fraction, left atrial diameter, the presence of flail leaflet, the presence of atrial fibrillations and the age of the subject | Within 30 days after the echo test

CONTACTS AND LOCATIONS:
Locations (1):
- RAMBAM health care center, Haifa, Israel